CLINICAL TRIAL: NCT04142983
Title: A Clinical Study of the Safety and Antibody Responses of Plasma Donors Vaccinated With a Licensed Tdap Vaccine
Brief Title: Tdap Vaccine Safety for Plasma Donors
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: GCAM Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GCAM-TET-01
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Results first posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Tetanus
MeSH Terms: conditions — Tetanus | interventions — adacel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): Participants will receive a single dose of Tdap vaccine (Adacel) every 3 months for a total of 5 immunizations over a period of 12 months.
  Interventions: Biological: Adacel

INTERVENTIONS:
Biological: Adacel — 0.5 mL, Intramuscular
  Other Names: Tdap Vaccine

SUMMARY:
This is a prospective, open label, single-arm, multi-center, Phase 1 study measuring the safety and tetanus antibody responses to Tdap vaccine administered to plasma donors every 3 months ±1 week for 12 months (5 vaccinations) with a 6 month follow-up after the last vaccination. After obtaining informed consent and screening for eligibility including plasmapheresis donor eligibility, subjects will have other baseline assessments performed and if eligible, will receive the scheduled vaccinations, will be assessed for adverse events (AEs) and have plasma samples collected for antibody titers each month thereafter for 11 months, and then at 1 and 6 months after the last vaccination. As these subjects are participating in a standard donor plasmapheresis donor program, assessments for donor eligibility and routine plasmapheresis will be performed; however, only the data specifically required to meet the objectives of this study will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ages 18 to 63 years
* Females of childbearing potential who agree to employ adequate birth control measures during the study
* Signed the informed consent form (ICF)
* Met all of the criteria required by GCAM to be a Normal Source Plasma donor
* Subject is not participating in any other immunization program

Exclusion Criteria:

* Subject is pregnant
* Subject has a condition or abnormality that in the opinion of the Investigator would compromise the safety of the subject or the quality of the data
* Subject has repeated reactions or hypersensitivity to components in the vaccine (e.g., thimerosal, latex, etc.)
* Subject has history of a severe reaction to any immunization
* Subject has a history of Guillain-Barré Syndrome
* The Investigator concludes that the anticipated vaccination site (deltoid area) is not suitable for AE assessment

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - GCAM Eagle Pass Center, Eagle Pass, Texas
  - GCAM Laredo Center, Laredo, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants between the ages of 18 to 63 years old were recruited from the Laredo, Texas area during February through May, 2020, without regard to ethnicity, race, or socioeconomic level. Standard recruiting practices such as IRB-approved flyers were used to recruit study volunteers
Pre-assignment Details: All participants were "Qualified Donors" who had been qualified for continued plasma donations in accordance with Donor Eligibility requirements found in 21 CFR 630.10 and 630.15, and Source Plasma regulations under 21 CRF 640, Subpart G. A total of 110 participants were consented and screened for eligibility. Ten of these did not meet eligibility criteria.
Groups:
- Tdap Vaccine: The vaccine was administered every 3 months ± 1 week for 12 months (5 vaccinations)
Period: Overall Study
Arm/Group | Tdap Vaccine
Started | 110
Treatment Population | 100
Completed | 11
Not Completed | 99
Not completed — Lost to Follow-up | 73
Not completed — Withdrawal by Subject | 10
Not completed — Physician Decision | 1
Not completed — Adverse Event | 1
Not completed — No longer eligible | 4
Not completed — Screen Failure | 10

BASELINE CHARACTERISTICS:
Arm/Group | Tdap Vaccine
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 100
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 100
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs are defined as an adverse event occurring after first study treatment. A serious TEAE was defined as an AE that resulted in any of the following outcomes: death; life-threatening; inpatient hospitalization or prolongation of hospitalization; persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, an important medical event that based on appropriate medical judgment may jeopardize the subject and may require medical or surgical intervention to prevent one of the aforementioned outcomes.
Time Frame: Up to 18 months
Population: Population included all enrolled participants who received at least one vaccination and had safety data.
Measure: Number; unit: participants
Groups:
- Tdap Vaccine: Tdap vaccine 0.5 mL administered intramuscularly on Day 0, Month 3, Month 6, Month 9 and Month 12.
Arm/Group | Tdap Vaccine
Number analyzed (Participants) | 100
participants
  Number of participants with at least one TEAE | 71
  Number of participants with at least one TEAE related to the study product | 42
  Number of participants with at least one serious TEAE | 0

2. Secondary Outcome: Anti-tetanus Antibody Titers in Participants Over Time
Description: Anti-tetanus antibody titer levels after each vaccination presented at geometric means (GeoMean) over time.
Time Frame: Baseline, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 7, Month 8, Month 9, Month 10, Month 11, Month 12, Month 13, Month 18
Population: Multiple participants dropped out of the study early. Missing data were documented in the protocol deviations and summary statistics to reflect the number of observations for which data were provided. No missing data were derived.
Measure: Geometric Mean (Standard Deviation); unit: Titers (IU/mL)
Arm/Group | Tdap Vaccine
Number analyzed (Participants) | 100
Titers (IU/mL)
  Screening | 1.2 (1.29)
  Month 1: number analyzed (Participants) | 74
  Month 1 | 13.2 (0.74)
  Month 2: number analyzed (Participants) | 72
  Month 2 | 8.1 (0.89)
  Month 3: number analyzed (Participants) | 70
  Month 3 | 5.6 (1.12)
  Month 4: number analyzed (Participants) | 68
  Month 4 | 9.0 (0.56)
  Month 5: number analyzed (Participants) | 64
  Month 5 | 5.9 (0.82)
  Month 6: number analyzed (Participants) | 62
  Month 6 | 4.8 (0.89)
  Month 7: number analyzed (Participants) | 55
  Month 7 | 7.8 (0.69)
  Month 8: number analyzed (Participants) | 51
  Month 8 | 5.8 (0.70)
  Month 9: number analyzed (Participants) | 49
  Month 9 | 4.5 (0.75)
  Month 10: number analyzed (Participants) | 44
  Month 10 | 7.7 (0.53)
  Month 11: number analyzed (Participants) | 42
  Month 11 | 5.1 (0.72)
  Month 12: number analyzed (Participants) | 34
  Month 12 | 4.2 (0.83)
  Month 13: number analyzed (Participants) | 39
  Month 13 | 6.3 (0.79)
  Month 18: number analyzed (Participants) | 1
  Month 18 | 5.0 (0.00)

3. Secondary Outcome: Number of Participants With Post Vaccination Anti-tetanus Antibody Range Levels
Description: The numbers and percentages of participants whose post vaccination antibody levels were <5 IU/mL; ≥5 IU/mL to 10 IU/mL; >10 IU/mL to 15 IU/mL; and, >15 IU/mL after each vaccination.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Tdap Vaccine
Number analyzed (Participants) | 100
Participants
  Screening: < 5 IU/mL | 88
  Screening: ≥ 5 to 10 IU/mL | 8
  Screening: ≥ 10 to 15 IU/mL | 4
  Screening: ≥ 15 IU/mL | 0
  Month 1: number analyzed (Participants) | 74
  Month 1: < 5 IU/mL | 4
  Month 1: ≥ 5 to 10 IU/mL | 22
  Month 1: ≥ 10 to 15 IU/mL | 12
  Month 1: ≥ 15 IU/mL | 36
  Month 2: number analyzed (Participants) | 72
  Month 2: < 5 IU/mL | 14
  Month 2: ≥ 5 to 10 IU/mL | 31
  Month 2: ≥ 10 to 15 IU/mL | 10
  Month 2: ≥ 15 IU/mL | 17
  Month 3: number analyzed (Participants) | 69
  Month 3: < 5 IU/mL | 23
  Month 3: ≥ 5 to 10 IU/mL | 29
  Month 3: ≥ 10 to 15 IU/mL | 9
  Month 3: ≥ 15 IU/mL | 8
  Month 4: number analyzed (Participants) | 68
  Month 4: < 5 IU/mL | 7
  Month 4: ≥ 5 to 10 IU/mL | 30
  Month 4: ≥ 10 to 15 IU/mL | 21
  Month 4: ≥ 15 IU/mL | 10
  Month 5: number analyzed (Participants) | 64
  Month 5: < 5 IU/mL | 15
  Month 5: ≥ 5 to 10 IU/mL | 34
  Month 5: ≥ 10 to 15 IU/mL | 12
  Month 5: ≥ 15 IU/mL | 3
  Month 6: number analyzed (Participants) | 62
  Month 6: < 5 IU/mL | 20
  Month 6: ≥ 5 to 10 IU/mL | 33
  Month 6: ≥ 10 to 15 IU/mL | 8
  Month 6: ≥ 15 IU/mL | 1
  Month 7: number analyzed (Participants) | 55
  Month 7: < 5 IU/mL | 8
  Month 7: ≥ 5 to 10 IU/mL | 29
  Month 7: ≥ 10 to 15 IU/mL | 10
  Month 7: ≥ 15 IU/mL | 8
  Month 8: number analyzed (Participants) | 51
  Month 8: < 5 IU/mL | 11
  Month 8: ≥ 5 to 10 IU/mL | 30
  Month 8: ≥ 10 to 15 IU/mL | 9
  Month 8: ≥ 15 IU/mL | 1
  Month 9: number analyzed (Participants) | 55
  Month 9: < 5 IU/mL | 20
  Month 9: ≥ 5 to 10 IU/mL | 26
  Month 9: ≥ 10 to 15 IU/mL | 3
  Month 9: ≥ 15 IU/mL | 6
  Month 10: number analyzed (Participants) | 44
  Month 10: < 5 IU/mL | 6
  Month 10: ≥ 5 to 10 IU/mL | 21
  Month 10: ≥ 10 to 15 IU/mL | 16
  Month 10: ≥ 15 IU/mL | 1
  Month 11: number analyzed (Participants) | 42
  Month 11: < 5 IU/mL | 15
  Month 11: ≥ 5 to 10 IU/mL | 23
  Month 11: ≥ 10 to 15 IU/mL | 4
  Month 11: ≥ 15 IU/mL | 0
  Month 12: number analyzed (Participants) | 34
  Month 12: < 5 IU/mL | 13
  Month 12: ≥ 5 to 10 IU/mL | 20
  Month 12: ≥ 10 to 15 IU/mL | 1
  Month 12: ≥ 15 IU/mL | 0
  Month 13: number analyzed (Participants) | 39
  Month 13: < 5 IU/mL | 5
  Month 13: ≥ 5 to 10 IU/mL | 27
  Month 13: ≥ 10 to 15 IU/mL | 6
  Month 13: ≥ 15 IU/mL | 1
  Month 18: number analyzed (Participants) | 1
  Month 18: < 5 IU/mL | 0
  Month 18: ≥ 5 to 10 IU/mL | 1
  Month 18: ≥ 10 to 15 IU/mL | 0
  Month 18: ≥ 15 IU/mL | 0

ADVERSE EVENTS:
Time Frame: 1 year, 6 months
Description: AEs and serious adverse events (SAEs) were collected starting with the initiation of the first study vaccination through study month 18, documented in the source records, and entered into the eCRFs using accepted medical terms and/or the diagnosis that accurately characterized the event.
Arm/Group | Tdap Vaccine
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 71/100
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tdap Vaccine (N=100)
Injection site pain (General disorders) | 37
Injection site bruising (General disorders) | 26
Injection site erythema (General disorders) | 14
Injection site induration (General disorders) | 8
Injection site swelling (General disorders) | 6
Red blood cells urine positive (Investigations) | 18
Urine leukocyte esterase positive (Investigations) | 17
Protein urine present (Investigations) | 14
Hemoglobin urine present (Investigations) | 11
Glucose urine present (Investigations) | 7
Urine ketone body present (Investigations) | 5
Headache (Nervous system disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-12-30): https://cdn.clinicaltrials.gov/large-docs/83/NCT04142983/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/83/NCT04142983/SAP_001.pdf